CLINICAL TRIAL: NCT00629278
Title: SHORT-HER: MULTICENTRIC RANDOMISED PHASE III TRIAL OF 2 DIFFERENT ADJUVANT CHEMOTHERAPY REGIMENS PLUS 3 VS 12 MONTHS OF TRASTUZUMAB IN HER2 POSITIVE BREAST CANCER PATIENTS
Brief Title: Combination Chemotherapy and Trastuzumab in Treating Women With Stage I, Stage II, or Stage III HER2-Positive Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: AOUMODENA-SHORT-HER; CDR0000584446 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2007-004326-25; EU-20825
Record Dates: First submitted 2008-03-04; First posted 2008-03-05 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Aromatase Inhibitors; Cyclophosphamide; Docetaxel; Doxorubicin; Epirubicin; Fluorouracil; Paclitaxel; Tamoxifen; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Biological: trastuzumab
Drug: aromatase inhibition therapy
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: paclitaxel
Drug: releasing hormone agonist therapy
Drug: tamoxifen citrate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known which regimen of combination chemotherapy given together with trastuzumab is most effective in treating breast cancer.

PURPOSE: This randomized phase III trial is comparing two different regimens of combination chemotherapy given together with trastuzumab to see how well they work in treating women with HER2-positive stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate if 3 months of trastuzumab (Herceptin®) administered according to the Finnish protocol (9-weekly administrations) is not inferior to 12 months (18 three-weekly administrations) in a standard chemotherapy protocol, in terms of disease-free survival, in patients with HER2-positive early breast cancer.
* To determine overall survival of patients treated with these regimens.

Secondary

* To determine the failure rate at 2 years, calculated as cumulative incidence of relapse, contralateral breast cancer (excluding in situ carcinoma), death for all causes, and treatment withdrawal due to toxicity of therapy.
* To determine the incidence of cardiac events (defined as decrease of ejection fraction (EF) over 15% from basal values, or decrease over 10% with EF absolute value below 50%, or symptomatic cardiac failure, or other cardiac side effects grade 2 or more according to NCI CTCAE v.3.

OUTLINE: This is a multicenter study. Patients are stratified according to nodal status (positive vs negative), hormone-receptor status (estrogen receptor-positive vs progesterone receptor-positive disease), and Regional Coordinating Center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (standard long-term adjuvant treatment-12 months): Patients receive chemotherapy comprising either doxorubicin hydrochloride IV and cyclophosphamide IV or epirubicin hydrochloride IV and cyclophosphamide IV on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients then receive paclitaxel IV over 3 hours or docetaxel* IV over 1 hour and concurrent trastuzumab (Herceptin®) IV over 90 minutes. Treatment repeats every 21 days for up to 4 courses.

NOTE: *Patients < 65 years old receive a higher dose of docetaxel and patients ≥ 65 years old receive a lower dose of docetaxel.

After completion of chemotherapy and concurrent trastuzumab, patients receive trastuzumab IV over 30-60 minutes as monotherapy every 21 days for up to 14 courses in the absence of disease progression or unacceptable toxicity.

* Arm II (experimental short-term adjuvant treatment-3 months): Patients receive docetaxel** IV on day 1. Treatment repeats every 21 days for up to 3 courses. Patients also receive trastuzumab IV over 30-60 minutes on day 1. Treatment repeats weekly for up to 9 weeks (9 doses).

Within 21 days after completion of docetaxel therapy, patients receive fluorouracil IV, epirubicin hydrochloride IV, and cyclophosphamide IV on day 1. Treatment repeats every 21 days for up to 3 courses.

NOTE: **Patients < 65 years old receive a higher dose of docetaxel and patients ≥ 65 years old receive a lower dose of docetaxel.

In both arms, patients treated with conservative surgery or those with more than 4 positive axillary nodes undergo radiotherapy within 8 weeks after completion of chemotherapy. Patients enrolled in arm I undergo radiotherapy concurrently with trastuzumab.

Patients with hormone receptor-positive tumor (i.e., estrogen receptor and/or progesterone receptor-positive tumor) also receive hormonal treatment after completion of chemotherapy. Patients enrolled in arm I receive hormonal therapy concurrently with trastuzumab.

Premenopausal patients receive monthly luteinizing-hormone releasing-hormone agonist for 2 years plus daily tamoxifen citrate for 5 years. Post-menopausal patients receive an aromatase inhibitor daily for 5 years.

After completion of study therapy, patients are followed for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of infiltrating primary breast cancer

  * Stage I-IIIA disease
  * Resected tumor with free margins (i.e., no neoplastic cells on the resected margin)

    * Must have node-negative sentinel node or complete axillary clearance

      * Axillary clearance required for micrometastasis (between 0.2 and 2 mm) in the sentinel node but not for isolated tumor cells
    * Treatment is scheduled to begin within 10 weeks from the date of surgery

      * Date of the last surgery will be taken into account for patients undergoing re-excision of positive margins or axillary lymph node dissection after positive sentinel node biopsy
* Node positivity or node negativity AND ≥ 1 of the following:

  * T > 2 cm
  * Grade 3
  * Presence of lymphovascular invasion
  * Ki 67 > 20%
  * Age 35 years
  * Hormone receptor negativity (<10%)
* HER2-positive tumor (3+ by IHC or FISH+ according to the American Society of Clinical Oncology guidelines [i.e., > 2.2; in case of polysomy, with ≥ 6 gene copies])
* Estrogen receptor-positive and/or progesterone receptor-positive disease

PATIENT CHARACTERISTICS:

* Female
* Pre- or postmenopausal status

  * Postmenopausal status defined by ≥ 1 of the following:

    * At least 60 years of age
    * Less than 60 years of age and amenorrheic for ≥ 12 months prior to day 1
    * Less than 60 years of age and amenorrheic for < 12 months prior to day 1 with luteinizing hormone and follicle-stimulating hormone values within postmenopausal range OR without a uterus
    * Prior bilateral oophorectomy
    * Prior radiation castration with amenorrhea for ≥ 6 months
* ECOG performance status 0-1
* Suitable for adjuvant chemotherapy
* WBC > 3,000/mcL
* ANC > 1,500/mcL
* Platelet count >100,000/mcL
* Total bilirubin normal
* AST and ALT 2.5 times upper limit of normal
* Creatinine normal
* Cardiac ejection fraction normal as measured by ECHO or MUGA scan
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study therapy
* No contraindication to anthracycline, cyclophosphamide, fluorouracil, paclitaxel, or trastuzumab (Herceptin®) treatment
* No uncontrolled intercurrent illness including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* See Patient Characteristics
* No prior chemotherapy, endocrine therapy, or radiotherapy
* No other concurrent investigational agents

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival
Overall survival

SECONDARY OUTCOMES:
Failure rate at 2 years due to relapse, death, or toxicity
Incidence of cardiac events as assessed by NCI CTCAE V3.0

CONTACTS AND LOCATIONS:
Overall Officials: Pier Franco Conte, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Modena
Locations (6):
- Italy (6):
  - Ospedale Santa Croce, Cuneo
  - Ospedale Civile di Ivrea, Ivrea
  - Azienda Ospedaliera - Universitaria di Modena, Modena
  - Piacenza Hospital, Piacenza
  - Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino, Turin
  - Ospedal San Andrea, Vercelli

REFERENCES:
- [Result] Guarneri V, Frassoldati A, Bruzzi P, D'Amico R, Belfiglio M, Molino A, Bertetto O, Cascinu S, Cognetti F, Di Leo A, Pronzato P, Crino L, Agostara B, Conte P. Multicentric, randomized phase III trial of two different adjuvant chemotherapy regimens plus three versus twelve months of trastuzumab in patients with HER2- positive breast cancer (Short-HER Trial; NCT00629278). Clin Breast Cancer. 2008 Oct;8(5):453-6. doi: 10.3816/CBC.2008.n.056. PMID 18952561
- [Derived] Conte P, Bisagni G, Piacentini F, Sarti S, Minichillo S, Anselmi E, Aieta M, Gebbia V, Schirone A, Musolino A, Garrone O, Beano A, Rimanti A, Giotta F, Turletti A, Miglietta F, Dieci MV, Vicini R, Balduzzi S, D'Amico R, Guarneri V. Nine-Week Versus One-Year Trastuzumab for Early Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer: 10-Year Update of the ShortHER Phase III Randomized Trial. J Clin Oncol. 2023 Nov 10;41(32):4976-4981. doi: 10.1200/JCO.23.00790. Epub 2023 Sep 25. PMID 37748109
- [Derived] Dieci MV, Bisagni G, Bartolini S, Frassoldati A, Vicini R, Balduzzi S, D'amico R, Conte P, Guarneri V. Type of adjuvant endocrine therapy and disease-free survival in patients with early HR-positive/HER2-positive BC: analysis from the phase III randomized ShortHER trial. NPJ Breast Cancer. 2023 Feb 4;9(1):6. doi: 10.1038/s41523-023-00509-2. PMID 36739285
- [Derived] Dieci MV, Bisagni G, Brandes AA, Frassoldati A, Cavanna L, Giotta F, Aieta M, Gebbia V, Musolino A, Garrone O, Donadio M, Rimanti A, Beano A, Zamagni C, Soto Parra H, Piacentini F, Danese S, Ferro A, Cagossi K, Sarti S, Gambaro AR, Romito S, Bazan V, Amaducci L, Moretti G, Foschini MP, Balduzzi S, Vicini R, D'Amico R, Griguolo G, Guarneri V, Conte PF. Validation of the AJCC prognostic stage for HER2-positive breast cancer in the ShortHER trial. BMC Med. 2019 Nov 21;17(1):207. doi: 10.1186/s12916-019-1445-z. PMID 31747948
- [Derived] Conte P, Frassoldati A, Bisagni G, Brandes AA, Donadio M, Garrone O, Piacentini F, Cavanna L, Giotta F, Aieta M, Gebbia V, Molino A, Musolino A, Ferro A, Maltoni R, Danese S, Zamagni C, Rimanti A, Cagossi K, Russo A, Pronzato P, Giovanardi F, Moretti G, Lombardo L, Schirone A, Beano A, Amaducci L, Bajardi EA, Vicini R, Balduzzi S, D'Amico R, Guarneri V. Nine weeks versus 1 year adjuvant trastuzumab in combination with chemotherapy: final results of the phase III randomized Short-HER studydouble dagger. Ann Oncol. 2018 Dec 1;29(12):2328-2333. doi: 10.1093/annonc/mdy414. PMID 30219886